CLINICAL TRIAL: NCT06428565
Title: Conventional Exercises Plan With or Without Laser Guided Feedback for Patients With Non-Specific Low Back Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MSRSW/Batch-Fall22/713
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low-level laser therapy (LLLT) or cold laser therapy (Experimental): uses low-level lasers or light-emitting diodes to stimulate cellular function and improve healing. Physiotherapy, sports medicine, and rehabilitation use it as a non-invasive, painless complement or adjuvant therapy
  Interventions: Diagnostic Test: Low-level laser therapy (LLLT) or cold laser therapy

INTERVENTIONS:
Diagnostic Test: Low-level laser therapy (LLLT) or cold laser therapy — Low-level laser therapy (LLLT) or cold laser therapy

SUMMARY:
Low back pain (LBP) is a significant health issue. It impacts a significant portion of the adult population, reaching up to 80%, and results in substantial healthcare and socioeconomic expenses. To find out what changes occurred after the application of two exercise modalities [Conventional Exercise (CE) and Laser-Guided Exercise (LGE)} and PNE on pain, pain pressure thresholds, disability, catastrophizing, kinesiophobia, and lumbar proprioception in subjects with NSCLBP.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female ages between 18 and 45 years (11).
* Patients diagnosed with nonspecific low back pain (11).
* patients with pain intensity of "3" or greater on numeric pain rating scale

Exclusion Criteria:

* Patients with neurological symptoms.
* Patients diagnosed with fatigue syndrome
* Females having pregnancy
* History of low back surgery

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
The Numeric Pain Rating Scale (NRS) | 12 Months
  it is a simple and widely used tool for measuring pain intensity. It consists of a horizontal line with 11 numbered points, ranging from 0 (no pain) to 10 (worst pain imaginable). Patients are asked to rate their pain by selecting the number that best describes their current pain intensity
The Oswestry Disability Index (ODI) | 12 months
  it is a patient-completed questionnaire used to measure the level of disability caused by low back pain. It is a widely used and validated tool in both research and clinical settings. Studies show high test-retest reliability of 0.90

CONTACTS AND LOCATIONS:
Locations (1):
- Hameed Latif Hospital Lahore, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No